CLINICAL TRIAL: NCT01295021
Title: A Non Interventional, Cross Sectional, Study on the Prevalence of Sympathetic Overactivity in Hypertensive Patients.
Brief Title: The Prevalence of Sympathetic Overactivity in Primary Hypertensive Patients.
Acronym: SORT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIN-DUM-2010/2
Record Dates: First submitted 2011-02-03; First posted 2011-02-14 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Essential Hypertension
Keywords: The prevalence of sympathetic overactivity in hypertensive patients.
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this NIS is to assess the prevalence of sympathetic overactivity in patients with newly diagnosed essential hypertension.

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed essential hypertension patients will be eligible for the study.
* Average of two or more systolic BP readings ≥ 140mmHg or diastolic BP readings ≥ 90mmHg

Exclusion Criteria:

* History of coronary artery disease
* History of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 1514 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of SO in newly diagnosed hypertensive patients | Visit 1-3: heart rate & Blood pressure, treatment presribed by physician. The interval between visit 1 and visit 2 is upto 4 weeks and interval between visit 2 & visit 3 is upto 4 weeks depending on Investigators discretion.

SECONDARY OUTCOMES:
Association of SO and heart rate. | Visits 1-3
Subjective symptoms noticed by the doctor. | 1st visit
To record the drugs used in the treatment of patients diagnosed with hypertension. | Visits 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Dr T.N.C. Padmanabhan, Principal Investigator — Dr. Padmanabhan Heart Clinic
Locations (97):
- India (97):
  - Research Site, Agartala
  - Research Site, Agra
  - Research Site, Ahmedabad
  - Research Site, Aligarh
  - Research Site, Ambattur
  - Research Site, Amritsar
  - Research Site, Aurangabad
  - Research Site, Bangalore
  - Research Site, Barelly
  - Research Site, Baroda
  - Research Site, Batanagar
  - Research Site, Beed
  - Research Site, Belagavi
  - Research Site, Bhagal
  - Research Site, Bhongi
  - Research Site, Bhopal
  - Research Site, Bhuj
  - Research Site, Burdwan
  - Research Site, Chandigarh
  - Research Site, Chennai
  - Research Site, Chomv
  - Research Site, Coimbatore
  - Research Site, Davangere
  - Research Site, Delhi
  - Research Site, Dhule
  - Research Site, Dombivali
  - Research Site, Ellisbridge
  - Research Site, Fariadad
  - Research Site, Faridabad
  - Research Site, Gandhinagar
  - Research Site, Ghatkopar East
  - Research Site, Ghaziabad
  - Research Site, Guntur
  - Research Site, Gūrgaon
  - Research Site, Gwalior
  - Research Site, Hanamkonda
  - Research Site, Hubli
  - Research Site, Hugli
  - Research Site, Hyderabad
  - Research Site, Indore
  - Research Site, Jabalpur
  - Research Site, Jaipur
  - Research Site, Jalandhar
  - Research Site, Jalgoon
  - Research Site, Kalaburagi
  - Research Site, Kanpur
  - Research Site, Karad
  - Research Site, Karīmnagar
  - Research Site, Kākināda
  - Research Site, Kolhāpur
  - Research Site, Kolkata
  - Research Site, Kulhapu
  - Research Site, Kumta
  - Research Site, Lucknow
  - Research Site, Ludhiana
  - Research Site, Madhyamgram
  - Research Site, Madurai
  - Research Site, Miroj
  - Research Site, Mohali
  - Research Site, Mozda
  - Research Site, Mrit Home
  - Research Site, Mulund East
  - Research Site, Mumbai
  - Research Site, Murshidābād
  - Research Site, Nadiād
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, Naugloi
  - Research Site, Navi Mumbai
  - Research Site, Nesul
  - Research Site, New Delhi
  - Research Site, New Panvel
  - Research Site, Newdelhi
  - Research Site, Nipāni
  - Research Site, Op Inchapur
  - Research Site, Panvel
  - Research Site, Parganas (Wb)
  - Research Site, Pālanpur
  - Research Site, Pune
  - Research Site, Raipur
  - Research Site, Rajkot
  - Research Site, Rajpur Sonarpur
  - Research Site, Sahibabad,Gzb
  - Research Site, Secenderabad
  - Research Site, Shakarpur
  - Research Site, Shimoga
  - Research Site, Sowcarpet
  - Research Site, Surat
  - Research Site, Thane
  - Research Site, Tirupati
  - Research Site, Ulhasnagar
  - Research Site, Vadodara
  - Research Site, Vijayawada
  - Research Site, Virār
  - Research Site, Visakhapatnam
  - Research Site, Vizag
  - Research Site, Warangal